CLINICAL TRIAL: NCT06357338
Title: Differential Expression and Potential Value of c-MYC in Non-invasive and Invasive Mammary Carcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Marwa Mahmoud Hassan (Other)
Collaborators: Qena Oncology Center (Other Government)
Responsible Party: Sponsor-Investigator, Marwa Mahmoud Hassan, resident doctor of pathologu, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-24-03-15MS
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Invasive Breast Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — formalin fixed, paraffin embedded tissue blocks of cases of mammary carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non invasive mammary carcinoma: 35 cases with non invasive breast cancer with low and high nuclear grades and co existing microfoci of invasion
  Interventions: Other: no intervention
- invasive mammary carcinoma: 35 cases of invasive breast cancer undergone MRM and classify them according grading, staging and luminal subtypes
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
Retrospective observational study to evaluate c-MYC expression in non invasive and invasive mammry carcinoma

DETAILED DESCRIPTION:
To correlate different levels of c-MYC expressions with variable clinical and pathological parameters of mammary carcinoma (such as patients' ages, tumor grading, staging, laterality, focality and nodal metastasis, co-existing in-situ components). This study will be carried out on archived formalin-fixed and paraffin embedded tissue blocks that were belonged to 70 women with breast lumps.

ELIGIBILITY:
Inclusion Criteria:

Specimens of Modified Radical Mastectomies from breast carcinoma patients

Exclusion Criteria:

* Cases with insufficient clinical data.

  * Tissue blocks of destroyed or insufficient material, unfit for diagnosis.
  * Cases who received pre-operative chemotherapy.

Min Age: 15 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: women with breast lumps administered to oncology center
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
role of c-MYC in breast cancer | 1 year
  difference between expression of c-MYC in non invasive and invasive mammary carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Alnashar, professor, Principal Investigator — Sohag University
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gao FY, Li XT, Xu K, Wang RT, Guan XX. c-MYC mediates the crosstalk between breast cancer cells and tumor microenvironment. Cell Commun Signal. 2023 Jan 31;21(1):28. doi: 10.1186/s12964-023-01043-1. PMID 36721232